CLINICAL TRIAL: NCT03662633
Title: Diagnosis Value of SEMA4C in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Hubei Cancer Hospital (Other); Qilu Hospital of Shandong University (Other); Wuhan Central Hospital (Other); Xiangyang Central Hospital (Other); The First People's Hospital of Jingzhou (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Clinical Professor, Tongji Hospital
Other Study IDs: 2018-TJ-BCD
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer group: Patients who have histologically confirmed new diagnosis of breast cancer are recruited.
  Interventions: Diagnostic Test: Breast cancer group
- Benign breast tumor group: Patients who have histologically confirmed new diagnosis of benign breast tumors are recruited.
  Interventions: Diagnostic Test: Benign breast tumor group

INTERVENTIONS:
Diagnostic Test: Breast cancer group — All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum SEMA4C levels were measured using a double antibody sandwich ELISA method using in-house SEMA4C detection kits.
  Groups: Breast cancer group
Diagnostic Test: Benign breast tumor group — All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum SEMA4C levels were measured using a double antibody sandwich ELISA method using in-house SEMA4C detection kits.
  Groups: Benign breast tumor group

SUMMARY:
Breast cancer remains the most common cancer in women worldwide. Early diagnosis can greatly improve the prognosis. To date, imaging examination is still the most important diagnostic and grading tool for breast cancer. Semaphorin4C (SEMA4C) has previously been identified as a highly expressed protein by breast cancer-associated lymphatic endothelial cells (LECs). The study is undertaken to evaluate the diagnostic efficiency of SEMA4C.

DETAILED DESCRIPTION:
Breast cancer remains the most common cancer in women worldwide, with approximately 1.68 million new cases, and 0.52 million deaths, annually. Meanwhile the incidence of breast cancer continues to increase. Early diagnosis and access to optimum treatment are crucial to reduce mortality associated with breast cancer. Currently, mammography and breast ultrasonography are essential for the detection and diagnosis of disease, and breast magnetic resonance imaging is the choice to estimate the extent of disease and guide appropriate treatment. However, there is no robust biomarkers for early detection of breast cancer.

Semaphorin4C (SEMA4C) has been previously identified as a highly expressed protein by breast cancer-associated lymphatic endothelial cells (LECs) using in situ laser capture microdissection of lymphatic vessels, followed by cDNA microarray analysis. Moreover, membrane-bound SEMA4C is cleaved by matrix metalloproteinase (MMPs) to release a soluble form of this protein. Therefore, this prospective project aims to assess the early diagnostic value of SEMA4C as a biomarker for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Receiving no treatment before diagnosis
* Establishing Diagnosis according to biopsy or surgery

Exclusion Criteria:

* Patients who are not mentally capable of giving written informed consent
* Clinical data missing
* Serum samples doesn't qualified
* Patients with a diagnosis of other severe acute or chronic medical conditions that may interfere with the interpretation of the study results

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants including patients with benign breast tumors and patients with breast cancer. All cases were confirmed histopathologically according to the WHO Classification of Tumors.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic potential of SEMA4C as a biomarker for breast cancer | At the time of inclusion
  Analyzing the predictive value of SEMA4C in the diagnosis of breast cancer.

SECONDARY OUTCOMES:
Serum SEMA4C, Mammography, breast US and MRI in comparison and combination to distinguish breast cancer from benign breast tumor | At the time of inclusion
  Compare and combine the diagnostic performances of Serum SEMA4C, traditional mammography, ultrasonography, and contrast-enhanced MR imaging in the assessment of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD, PhD, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wei JC, Yang J, Liu D, Wu MF, Qiao L, Wang JN, Ma QF, Zeng Z, Ye SM, Guo ES, Jiang XF, You LY, Chen Y, Zhou L, Huang XY, Zhu T, Meng L, Zhou JF, Feng ZH, Ma D, Gao QL. Tumor-associated Lymphatic Endothelial Cells Promote Lymphatic Metastasis By Highly Expressing and Secreting SEMA4C. Clin Cancer Res. 2017 Jan 1;23(1):214-224. doi: 10.1158/1078-0432.CCR-16-0741. Epub 2016 Jul 8. PMID 27401250
- [Background] Gurrapu S, Pupo E, Franzolin G, Lanzetti L, Tamagnone L. Sema4C/PlexinB2 signaling controls breast cancer cell growth, hormonal dependence and tumorigenic potential. Cell Death Differ. 2018 Jul;25(7):1259-1275. doi: 10.1038/s41418-018-0097-4. Epub 2018 Mar 19. PMID 29555978